CLINICAL TRIAL: NCT06994624
Title: Clinical and Biochemical Effects of a Defined Plant-Based Diet on Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Johnsie and Aubary Montgomery Institute of Medical Education and Research (Other)
Responsible Party: Principal Investigator, Rami Najjar, Postdoctoral Fellow, Georgia State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20212729
Record Dates: First submitted 2025-04-25; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will consume a defined, plant-based diet (PBD) and receive standard medical care. Subjects will consume their diets for 42-days and all food will be provided, although subjects are free to consume ad libitum within their assigned dietary protocols. Supplement use will be discontinued unless clinically indicated. As previously described, participants consuming the DPBD will consume foods within a proprietary food classification system consisting of levels 0-4b.26 These include raw fruits, berries, vegetables, oats, buckwheat, seeds and avocado. Excluded for consumption are cooked foods, animal products, free oils, soda, alcohol and coffee. The Garden Kitchen™ (Houston, TX) will provide food for subjects consuming the PBD. Dietary intake will be monitored via a 24-hour dietary recall at baseline and at day 28. All subjects will be monitored with weekly telephone or office visits by a clinical team member.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant-based diet (Experimental): This group will consumed a plant-based diet for 6 weeks.
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — A plant-based diet

SUMMARY:
A plant-based diet will be utilized in the treatment of coronary artery disease.

DETAILED DESCRIPTION:
Study population Men and women who have been diagnosed with coronary artery disease (CAD) at Montgomery Heart & Wellness Clinic in Houston, TX will be recruited to participate in this randomized study. Subjects will be recruited through flyers and social media advertisements. Also, subjects should currently follow a standard western diet. Exclusion criteria include the following: current tobacco use, excessive alcohol use (defined as >2 glasses of wine or alcohol equivalent per day for men or >1 glass of wine or alcohol equivalent for women), a current cancer diagnosis, an ongoing clinically defined infection, ≥ stage 3 kidney, current pregnancy or lactation, and prior hospitalization within past 6 months.

Dietary protocol Patients will consume a defined, plant-based diet (PBD) and receive standard medical care. Subjects will consume their diets for 42-days and all food will be provided, although subjects are free to consume ad libitum within their assigned dietary protocols. Supplement use will be discontinued unless clinically indicated. As previously described, participants consuming the DPBD will consume foods within a proprietary food classification system consisting of levels 0-4b.26 These include raw fruits, berries, vegetables, oats, buckwheat, seeds and avocado. Excluded for consumption are cooked foods, animal products, free oils, soda, alcohol and coffee. The Garden Kitchen™ (Houston, TX) will provide food for subjects consuming the PBD. Dietary intake will be monitored via a 24-hour dietary recall at baseline and at day 28. All subjects will be monitored with weekly telephone or office visits by a clinical team member.

Assessment of arrhythmias To assess any arrhythmias, a carnation ambulatory telemetric monitor, a non-invasive patch placed over the sternum, will monitor cardiac rhythms for 14-days prior to dietary initiation and 14 days after the 4 weeks are complete. The percent arrhythmic burden will be automatically determined by the monitor, characterized by rapid, irregular fibrillatory waves that vary in size, shape and timing.

Biochemical analysis Blood will be collected after a 12-h fast. A standard lipid panel measuring total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol and triglycerides will be obtained at baseline and 28 days. In addition, inflammatory biomarkers, such as hs-CRP will also be obtained. These biomarkers will be assessed by Quest Diagnostics (Secaucus, NJ) Additional blood will be collected in red-capped venous blood collection tubes intended for serum collection. Blood will allowed to sit at room temperature for 30 min, then spun down at 5,000 RPM for 10. Blood tubes will be shipped overnight to Georgia State University (Atlanta, GA) for serum analysis and cell culture experiments. Of particular interest are antioxidant enzymes superoxide dismutase (SOD), glutathione peroxidase (GPx1) and catalase. Additionally, inflammatory cytokine concentrations of interleukin (IL)-6, IL-1β and tumor necrosis factor (TNF)-a will be assessed with enzyme-linked immunosorbent assay (ELISA). Nitric oxide and myeloperoxidase (MPO) will also be measured in the serum, indicative of endothelial and systemic oxidative stress. Commercially available kits Superoxide Dismutase Assay Kit, Nitrate/Nitrite Colorimetric Assay Kit, Catalase Activity Assay Kit, TNF-α (human) ELISA Kit, Interleukin-6 (human) ELISA Kit, Interleukin-1β (human) ELISA Kit, Myeloperoxidase (MPO) Activity Assay Kit and Glutathione Peroxidase Assay Kit (Cayman Chemical, Ann Arbor, MI) be used to determine the concentrations of these proteins and molecules. Human cardiomyocytes and aortic endothelial cells purchased from PromoCell (Heidelberg, Germany) will be treated with isolated serum at baseline and at 4 weeks. After 24 h incubation, cells will be collected for protein analysis, gene analysis and for morphological observations.

Endothelial function Endothelial dysfunction is tightly tied with increased reactive oxygen species and systemic inflammation, and normal endothelial function is compromised in those with CAD. Thus, assessing changes in endothelial dysfunction is prudent. [10] Endothelial-dependent vasodilation will be measured using the reactive hyperemia index (RHI) at baseline and 28 days. Participants will be asked to fast overnight (10-12 h) and refrain from all medications (including aspirin), alcohol, and caffeine for at least 24 h before reporting to the study site in the morning. Upon arrival to the study site, appropriate-sized BP and two probes will be also placed on the participant's arms and index finger of both hands, respectively. The peripheral arterial tone (PAT) signal will be measured before and after hyperemia, blood flow occlusion using a non-invasive plethysmographic method (Endo-PAT 2000, Itamar Medical Ltd). Next, BP cuff will be inflated to 60 mmHg above SBP or 200mmHg, whichever is higher, for 5 min. The cuff will then be deflated to induce reactive hyperemia and PAT signal will be recorded for another 5 min. The RHI, post-to-pre-occlusion PAT signal ratio in the occluded arm, relative to the same ratio in the control arm, and corrected for baseline vascular tone, will be calculated.

Statistical analysis Based on power analysis utilizing our preliminary data, a sample size of 15 subjects per group is sufficient to demonstrate significance between groups. A P-value = 0.05 will be deemed significant. A mixed-effect analysis of variance model will be performed followed by post-hoc analysis to find differences between groups and across time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with coronary artery disease (based on current EKG or prior diagnosis)
* New patient

Exclusion Criteria:

* Current tobacco use

  ->2 glasses of wine for woman, >1 glass for men
* Current cancer diagnosis
* An ongoing clinically defined infection
* eGFR < 30
* Pregnancy
* Lactation
* Prior hospitalization within past 6 months
* Unstable angina
* Heart catheterization within past 6 months
* Cardiac perfusion study past 6 months
* Have not been on any form of a plant-based diet previously

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Improved endothelial function via reactive hyperemia index (RHI) | enrollment and at week 4
  Peripheral microvascular function will be measured by PAT plethysmographic device (EndoPAT, Itamar®). The device consists of a finger probe with a transducer to assess digital volume changes accompanying pulse-waves. An inflatable cuff is placed on one arm (test arm), while amplitudes are recorded from the test arm and the contralateral control arm. Reactive hyperemia index (RHI) is obtained by the following: 5 minutes of baseline amplitude signal detection, 5 minutes of arterial occlusion by suprasystolic cuff inflation, and then 6 min of post-occlusion amplitude signal detection. RHI is a unit-less measure calculated as a ratio of hyperemic to baseline flow signal. It takes into account the baseline signal and adjusts it to the changes in the contralateral arm

SECONDARY OUTCOMES:
Arrythmia assessment | Weeks 1-2 and weeks 7-8.
  Ambulatory telemetric monitor will be used for a 14-day period to assess abnormal incidents of QRS complex waves. These abnormal incidents will be counted and quantified. This is an external devise that uses ECG electrodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Montgomery Heart & Wellness Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified medical data, including endothelial function and telemetry data.

REFERENCES:
- [Background] Najjar RS, Moore CE, Montgomery BD. A defined, plant-based diet utilized in an outpatient cardiovascular clinic effectively treats hypercholesterolemia and hypertension and reduces medications. Clin Cardiol. 2018 Mar;41(3):307-313. doi: 10.1002/clc.22863. Epub 2018 Mar 25. PMID 29575002